CLINICAL TRIAL: NCT01925651
Title: Randomized Clinical Trial of the Impact of the Use of Bolus in the Treatment of Post Mastectomy Radiotherapy for Breast Cancer
Brief Title: Clinical Trial of The Use of Bolus in Post Mastectomy Irradiation in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Principal Investigator, Lucas Gomes Sapienza, Medical Doctor, AC Camargo Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC-B 01
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Radiodermatitis
Keywords: Post Mastectomy Radiotherapy; Breast Cancer; Bolus; Radiodermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard Risk - No bolus (Other): No Bolus
  Interventions: Radiation: No Bolus
- Standard Risk - Alternate Bolus (Other): Alternate 5mm Bolus
  Interventions: Radiation: Alternate Bolus
- High Risk - Alternate Bolus (Other): Alternate 5mm Bolus
  Interventions: Radiation: Alternate Bolus
- High Risk - Continuous bolus (Other): Continuous 5mm bolus
  Interventions: Radiation: Continuous Bolus

INTERVENTIONS:
Radiation: No Bolus — no bolus use
  Arms: Standard Risk - No bolus
Radiation: Alternate Bolus — 0.5cm bolus use in alternate days
  Arms: High Risk - Alternate Bolus; Standard Risk - Alternate Bolus
Radiation: Continuous Bolus — 0.5 cm bolus use in continuous days
  Arms: High Risk - Continuous bolus

SUMMARY:
The aim of this study is to evaluate the impact of adding bolus in adjuvant radiotherapy after mastectomy, in relation to the time of treatment interruption and acute effects. This study evaluates whether there is an increase in treatment time with the addition of the bolus, which can overshadow the benefit of increased dose to the skin and subcutaneous tissue. The patients will continue to be followed for oncologic outcomes, focusing on chest wall local control.

DETAILED DESCRIPTION:
Rational:

* The use of high-energy photons (6 MeV) creates a characteristic skin-sparing effect, which can generate a region of low-dose subcutaneous tissue.
* The subcutaneous tissue is a possible area of clinical failure in the chest wall after mastectomy for breast cancer.
* To optimize treatment, it is used a bio-equivalent material to increase the surface dose.
* This dose increase may be accompanied by greater skin reaction, making it necessary to temporarily discontinue treatment to recover radiodermatitis.
* The total treatment time is a determinant of tumor control in the treatment of cancer with radiation.

Description:

* This study aims to evaluate whether different intensities of application of the bolus correlate with greater likelihood of treatment discontinuation.
* This will be a single blind randomised controlled trial. The target population comprises patients with indication of post mastectomy radiation (PMRT).
* The patients will be divided into two groups: one with higher risk of recurrence in subcutaneous, which will be randomized to use 0.5cm bolus every other day or on consecutive days, and one lower risk group, which will be randomized to use bolus 0.5cm on alternate days or do not use bolus. The group with high risk is defined as patients with clinical or pathological tumor invasion of skin. The others will be considered standard risk.
* Randomization will be made so that each group has the same proportion of patients with high body mass index (> / = 30 kg/m2), as this may be a factor in worsening radiodermatitis.
* The patients will be followed during treatment and will be evaluated weekly for the radiodermatitis, interruption time of treatment for recovery from the acute effects and expenditures for local care. The evaluation will be done blindly (without knowledge of the utilization of bolus) by trained nurses in the management of radiodermatitis. After treatment, patients will continue to be followed for oncologic outcomes, focusing on chest wall local control.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing mastectomy with or without reconstruction of early breast
* breast malignancy histologically proven
* protocol addended to allow inclusion of men that meet all inclusion criteria

Exclusion Criteria:

* Karnofsky Performance Scale (KPS) <70%
* Concomitant chemotherapy (only permitted or hormone therapy molecular-targeted)
* Prior ipsilateral thoracic / cervical irradiation
* Proven metastatic disease (excluded from oncologic outcomes analyses)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Acute radiodermatitis | participants will be followed for the duration of radiotherapy, an expected average of 6 weeks
  Radiation Therapy Oncology Group (RTOG) grading system Common Terminology Criteria for Adverse Events (CTCAE) - v4.0

SECONDARY OUTCOMES:
Interruption Time | participants will be followed for the duration of radiotherapy, an expected average of 6 weeks
  Treatment Interruption time due to radiodermatitis

OTHER OUTCOMES:
Local Care Costs | participants will be followed for the duration of radiotherapy, an expected average of 6 weeks
  Local Care Costs with radiodermatitis
Local Control | From date of randomization until the date of first documented local progression in the chest wall or date of death from any cause, whichever came first, assessed up to 100 months
  local control in the chest wall assessed by physical examination and complementary exams.
Metastasis-Free Interval | From date of randomization until the date of first documented distant progression or date of death from any cause, whichever came first, assessed up to 100 months
  Metastasis-Free Interval (following departmental post-treatment surveillance visits routine).
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival (following departmental post-treatment surveillance visits routine).

CONTACTS AND LOCATIONS:
Overall Officials: Lucas G Sapienza, MD, PhD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil